CLINICAL TRIAL: NCT03278119
Title: Sleep Aging and Risk for Alzheimer's Resubmission 2.0
Brief Title: Sleep Aging and Risk for Alzheimer's 2.0
Acronym: SARA
Status: Active, not recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 17-01005; R01AG056031 (NIH)
Record Dates: First submitted 2017-09-07; First posted 2017-09-11 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease; Sleep Apnea
MeSH Terms: conditions — Alzheimer Disease; Sleep Apnea Syndromes | interventions — Positron-Emission Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sleep Apnea: Overall 56
  * both male and female
  * age group 55 to 75 years, having mild to severe obstructive sleep apnea
  * in good general health with no significant comorbidities
  * Located for the most part in boroughs of New York City
  Interventions: Diagnostic Test: PET Scan and nocturnal polysomnography
- No Sleep Apnea: Overall 56
  * both male and female
  * age group 55 to 75 years, without OSA
  * in good general health with no significant comorbidities
  * Located for the most part in boroughs of New York City
  Interventions: Diagnostic Test: PET Scan and nocturnal polysomnography

INTERVENTIONS:
Diagnostic Test: PET Scan and nocturnal polysomnography — Amyloid PET scans will be used to assess amyloid burden in the brain, and nocturnal polysomnography will be used to assess sleep and cardiopulmonary variables

SUMMARY:
Age-related sleep changes and common sleep disorders like obstructive sleep apnea (OSA) may increase amyloid burden and represent risk factors for cognitive decline in the elderly. We will directly interrogate the brain using a 2-night nocturnal polysomnography (NPSG) and amyloid deposition using C-PiB PET/MR both at baseline and at the 24-month follow-up. This study has the potential to identify the mechanisms by which age-related sleep changes contribute to AD neurodegeneration in cognitively normal elderly, the group that could profit the most from sleep preventive strategies.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, an individual must meet all of the following criteria:

* Male and female subjects with normal cognition and 55-75 years.
* Within normal limits on neurological and psychiatric examinations. All subjects enrolled will have a CDR=0.
* All subjects will have had a minimum of 12 years of education. Among minority subjects >80% of the elderly individuals coming to the NYU-ADC meet this criterion. The education restriction reduces performance variance on cognitive test measures and improves the sensitivity for detecting pathology and disease progression using the robust norms available at NYU. Given most subjects will meet this criterion we do not consider this a major selection bias or generalization limitation for this study.
* An informed family member or life-partner (preferably bed-partner) will be interviewed to confirm the reliability of the subject interview.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* History of brain tumor, MRI evidence of brain damage or brain disease including significant trauma, hydrocephalus, seizures, mental retardation or other serious neurological disorder (e.g. Parkinson's disease or other movement disorders).
* Significant history of alcoholism or drug abuse.
* History of psychiatric illness (e.g., schizophrenia, bipolar, PTSD, or life-long history of major depression).
* Geriatric Depression Scale (short form)>6.
* Insulin dependent diabetes.
* Evidence of clinically relevant cardiac, pulmonary, endocrine or hematological conditions.
* Physical impairment of such severity as to adversely affect the validity of psychological testing.
* Any prosthetic devices (e.g., pacemaker or surgical clips) that constitutes a hazard for MRI imaging.
* Medications affecting cognition: Narcotic analgesics, chronic use of medications with anticholinergic activity, anti-Parkinsonian medications (carbidopa/levodopa, amantadine, bromocriptine, selegiline). Others: amphetamines, amphetamine-like compounds, appetite suppressants, phenothiazines, reserpine, buspirone, clonidine, disulfiram, guanethidine, MAO inhibitors, theophylline, tricyclic antidepressants, salicylates, cholinesterase inhibitors and memantine.
* History of a first-degree family member with early onset (age <60 years) dementia.
* Irregular sleep-wake rhythms (based on the actigraphy recordings) or severe OSA (AHI4%≥30).
* Chronic use of antidepressants and melatonin are allowed.
* Excessive daytimes sleepiness (Epworth Sleepiness Scale >10) or history of CVE (arrhythmias, heart valve disease, cardiomyopathy, carotid or coronary artery disease and chest pain) will not be allowed in the OSA groups.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 112 subjects with normal sleep breathing (non-OSA) or mild to moderate OSA (AHI4%<30).
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Establishing how mild-to-moderate OSA increases AD risk will inform novel preventive therapies for AD. | 2.5 years

SECONDARY OUTCOMES:
Establishing that SWS quality is associated with longitudinal amyloid deposition will identify a key mechanism by which age increases AD risk. | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Osorio, MD, Principal Investigator — New York Langone Medical Center
Locations (1):
- Healthy Brain Aging and Sleep Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided